CLINICAL TRIAL: NCT05664529
Title: Evaluation of Mother-Child Interactions During Feeding in Toddlers
Brief Title: Mother-Child Interactions During Feeding
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2022.585
Record Dates: First submitted 2022-12-16; First posted 2022-12-23 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Feeding Disorders; Mother-Child Relations; Feeding; Disorder, Nonorganic Origin, in (Very Young) Child; Postpartum Depression
Keywords: child; feeding disorders; maternal depression
MeSH Terms: conditions — Feeding and Eating Disorders; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy children aged 6-36 months: 120 healthy children with or without any feeding difficulties reported by the mothers will be included. A 20-minute videotaped feeding session will be evaluated by Chatoor Feeding Scale to examine mother-infant relationship during feeding.
  Interventions: Diagnostic Test: Chatoor Feeding Scale

INTERVENTIONS:
Diagnostic Test: Chatoor Feeding Scale — Chatoor Feeding Scale will be used to evaluate mother infant relationship during feeding. Mothers will be asked to record a natural feeding session at home by video. The videos will be sent to the investigators by the parents. The first 20 minutes of the video will be evaluated for scoring.

SUMMARY:
The feeding process is based on a mutual relationship and interaction, as it takes place with the active participation of the child and the parent. Feeding problems are among the most common behavioral problems in early childhood. Inappropriate eating habits can cause growth retardation, unhealthy food preferences, and obesity. Parent-child interaction during feeding is particularly important in developing healthy feeding behavior.

The aim of this study is to evaluate the interaction between mother and child during feeding, by using the Feeding Scale in Turkish children aged 6-36 months.

A cross sectional, observational study will be conducted to explore mother-child relationship during feeding period by using Chatoor Feeding Scale.

DETAILED DESCRIPTION:
Healthy feeding practices are particularly important in the early childhood due to rapid growth. Between 25 and 40% of healthy infants, and 80% of infants with a health problem have feeding problems. Almost 50% of mothers complain that at least one of their children eats inadequate amount of food. Feeding problems in early childhood includes prolonged, disruptive and stressful mealtimes, food refusal, lack of appropriate independent feeding, nocturnal eating, distraction to increase intake and prolonged breast or bottle feeding.

Eating behavior is a social process, also have a biological aspect. After excluding organic causes of feeding problems, family's attitude, roles and expectations must be examined. The determination of family responsibilities, feeding habits, life styles, perceptions and concerns can be guidance for understanding of feeding difficulties.

Mothers are primarily responsible for child care and feeding process traditionally. Many factors such as mother's knowledge about feeding, cultural believes, workload, media effect, psychological symptoms, child's temperament, time spent together are important points on feeding process.

Verbal and non-verbal communication methods can be learned by the observation of family members at the mealtime. Eating disorder of the child and depression of the mother can be related to each other. Anxiety level, anger, lack of empathy and also child's irritability and negative mood can disturb interaction during feeding. As a result of unresponsiveness to child's eating skills and signals, food refusal can be seen. Oppressive and restrictive style can trigger different pathological conditions related with feeding process.

Mother-child interactions in the etiology of feeding disorders has been investigated by a series of studies. The initial studies used nonorganic failure to thrive (NOFTT) as a diagnosis for children younger than 3 years of age who were unable to gain weight inadequately due to behavioral problems related to feeding. Some other "behavioral style" studies also suggested to use Mealtime Observation Schedule, DSM-IV (Diagnostic and Statistical Manual) Criteria, Diagnostic Classification of Mental Health and Developmental Disorders of Infancy and Early Childhood-Revised Edition (DC:0-3R) as a diagnostic category of feeding disorder of infancy or early childhood. Feeding Scale developed by Chatoor is a useful tool to evaluate mother-child interactions during feeding.

This study is designed to observe and evaluate the relationship between child and mother during feeding at home in the transition to complementary feeding.

Our primary objective is to examine the mother infant relationship by using the Feeding Scale in infants aged 6 to 36 months. Parents of children aged between 6 and 36 months examined in Marmara University Hospital Pediatrics outpatient clinics will be informed about the study, and informed consent will be obtained on a voluntary basis if they wish to participate. A home video record during a regular mealtime will be requested from mothers. Mother will be instructed to feed the baby as she always does and record the mealtime by video or phone without distracting the baby. If the child still wishes to continue feeding after 20 minutes, the video recording will be allowed to continue until the mother ends the mealtime. However, in the scale evaluation, only the interactions in the first 20 minutes will be scored.

It is aimed to divide the intended audience into age groups according to developmental age groups. Therefore, a total of 120 mother-infant couples (dyads) including 30 children between 6-12 months, 30 children between 12-18 months, 30 children between 18-24 months and 30 children between 24-36 months will be targeted to include in the study.

Secondary objectives are to examine other factors affecting mother-infant relationship during feeding, such as neurodevelopment (assessed by Denver II), maternal anxiety (Generalized Anxiety Disorder-7), maternal depression (Edinburgh postpartum depression scale), postpartum bonding (The Postpartum Bonding Questionnaire) and baby sleep (Brief infant sleep questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* healthy children 6-36 months of age from outpatient pediatric clinics with parents willing to participate into the study

Exclusion Criteria:

* Children with chronic diseases

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy children aged between 6-36 months and their parents
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Feeding Scale scores | baseline
  Chatoor Feeding Scale will be used to evaluate mother-infant relationship during feeding. 20-minute at home videotaped feeding session will be evaluated. The Feeding Scale is composed of 46 items scored on a 4-point Likert scale (from 0 o 3) of how often and how intensely each of the behaviors occurred. The scale is composed of five subscales: Factor I (Dyadic Reciprocity) was a positive behavior while the remaining four factors (Dyadic Conflict, Talk and distraction, Struggle for Control, Maternal Non- Contingency) reflected negative behaviors. Unit scores were summed to produce factor scores and a high score for all factors reflect higher amounts of the behavior.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder questionnaire-7 scores of mothers | baseline
  It is a seven item scale developed to screen for anxiety in general in primary care settings. The questionnaire score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. Cut off score for Turkish validation has been set at 8.
Edinburgh postnatal depression scale (EPDS) scores of mothers | baseline
  Maternal depression will be measured by Edinburgh postnatal depression scale (EPDS). This is a 10-item self-administered scale (scores of 0,1,2 and 3), developed for detection of symptoms of psychosocial distress during pregnancy and in the postnatal period. The tool has been validated to Turkish. A score of >12 's at as the cut off point.
The Postpartum Bonding Questionnaire | baseline
  The scale consists of 25 items, with four factors. The first factor was labelled general emotional factor, the second anger towards and rejection of baby; the third infant-focus anxiety; and the fourth, risk of abuse. The scale was found reliable in Turkish.
Parental report of infant sleep patterns using the Brief Infant Sleep Questionnaire | baseline
  Infant sleep parameters will be measured by Expanded-Brief Infant Sleep Questionnaire (BISQ) : BISQ is a screening questionnaire for sleep in infants and young children. Variables include nocturnal sleep duration, daytime sleep duration, number of night wakenings, duration of night time wakefulness, nocturnal sleep onset time, settling time, method of falling asleep, location of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Perran Boran, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Requests for wider sharing of data (for example in response to information on the, Marmara University webpages and in publications about the study and willingness to share), will be addressed on a case-by-case basis. Any data sharing request will be made to investigators through a pre-defined data requisition form. This form will contain information about the applicant, institution, purpose of data request, study objectives, ethical clearance of the study, etc. Once a request has been made the data governance body will discuss if that request was appropriate and meets the criteria set by the participating centres; data will be released following signing of the data sharing agreement. The data will be stored on the Marmara University servers and not be deposited in any 'community' database.

REFERENCES:
- [Background] Chatoor I, Hommel S, Sechi C, Lucarelli L. DEVELOPMENT OF THE PARENT-CHILD PLAY SCALE FOR USE IN CHILDREN WITH FEEDING DISORDERS. Infant Ment Health J. 2018 Mar;39(2):153-169. doi: 10.1002/imhj.21702. Epub 2018 Feb 27. PMID 29485687
- [Background] Reisz S, Aviles AI, Messina S, Duschinsky R, Jacobvitz D, Hazen N. Fathers' attachment representations and infant feeding practices. Appetite. 2019 Nov 1;142:104374. doi: 10.1016/j.appet.2019.104374. Epub 2019 Jul 22. PMID 31344420
- [Background] Wendt V, Bergmann S, Herfurth-Majstorovic K, Keitel-Korndorfer A, von Klitzing K, Klein AM. Parent-child interaction during feeding or joint eating in parents of different weights. Eat Behav. 2015 Aug;18:131-6. doi: 10.1016/j.eatbeh.2015.04.007. Epub 2015 May 10. PMID 26051882
- [Background] Cerniglia L, Cimino S, Ballarotto G. Mother-child and father-child interaction with their 24-month-old children during feeding, considering paternal involvement and the child's temperament in a community sample. Infant Ment Health J. 2014 Sep-Oct;35(5):473-81. doi: 10.1002/imhj.21466. Epub 2014 Aug 13. PMID 25798497
- [Background] Chatoor I, Sechi C, Vismara L, Lucarelli L. A cross-sectional study of father-daughter/son interactions from 1 Month to 3 years of age with the feeding and play scales: Exploring the psychometric properties. Appetite. 2022 Jan 1;168:105671. doi: 10.1016/j.appet.2021.105671. Epub 2021 Sep 1. PMID 34481013